CLINICAL TRIAL: NCT02601326
Title: Laparoscopic Ventral Mesh Rectopexy Versus Delorme's Operation in Management of Complete Rectal Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mansourau24
Record Dates: First submitted 2015-10-28; First posted 2015-11-10 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2015-11

CONDITIONS: Complete Rectal Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic ventral mesh Rectopexy (Active Comparator): Fixation of the rectum to the sacrum using laparoscopy and mesh
  Interventions: Procedure: Laparoscopic ventral mesh Rectopexy
- delorme's procedure (Active Comparator): excision of excess rectal mucosa under spinal anesthesia then plication of the rectal muscles with vicryl 2/0 sutures
  Interventions: Procedure: Delorme's procedure

INTERVENTIONS:
Procedure: Laparoscopic ventral mesh Rectopexy — Laparoscopic fixation of rectum to sacral promontory using mesh
  Arms: Laparoscopic ventral mesh Rectopexy
Procedure: Delorme's procedure — Transanal excision of rectal mucosa and plication of muscle layer
  Arms: delorme's procedure

SUMMARY:
A comparative randomized study between laparoscopic ventral mesh Rectopexy and Delorme's procedure in treatment of complete rectal prolapse to ass both efficacy and complications

DETAILED DESCRIPTION:
A comparative randomized study between laparoscopic ventral mesh Rectopexy and Delorme's procedure in treatment of complete rectal prolapse to ass both efficacy and complications.

Follow up is scheduled for 18 months to evaluate recurrence, continence state and complications

ELIGIBILITY:
Inclusion Criteria:

* patients with complete rectal prolapse

Exclusion Criteria:

* patients who underwent previous surgery for complete rectal prolapse
* patients unfit for surgery
* patients with associated colorectal diseases or pathology

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Recurrence of the condition | 18 month
  Measured by counting the number of patients with recurrence of rectal prolapse

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Emile, M.D, Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided